CLINICAL TRIAL: NCT06874075
Title: Psychiatric Disorders in Child and Adolescent Offspring of Parents with Schizophrenia and Bipolar Disorders.
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Alshimaa Mohamed Saad, Assistant lecture, Assiut University
Other Study IDs: psychiatric marriage outcome
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-03

CONDITIONS: Mood Disorders; Schizophrenia Disorders
Keywords: bipolar; schizophrenia
MeSH Terms: conditions — Mood Disorders; Schizophrenia

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Offspring of parents with bipolar disorder (BD) and schizophrenia (SZ) are vulnerable and at high risk for these disorders. Despite the fact that positive family history of SZ or BD is the strongest predictor for the development of these severe mental illnesses, there is limited evidence assessing young adults of SZ and BP simultaneously with lack of detailed handling of similarities in risk and developmental trajectories during adolescence

DETAILED DESCRIPTION:
Offspring of parents with bipolar disorder (BD) and schizophrenia (SZ) are vulnerable and at high risk for these disorders. Despite the fact that positive family history of SZ or BD is the strongest predictor for the development of these severe mental illnesses, there is limited evidence assessing young adults of SZ and BP simultaneously with lack of detailed handling of similarities in risk and developmental trajectories during adolescence [1, 2]. SZ and BP are thought to share a common pathophysiological basis due to advances in the field of molecular genetics, which have yielded overlapping findings between the two disorders [3, 4]. The psychopathological base during adolescence is influenced by neurodevelopmental deviation prior to clinical onset of many severe mental illnesses [5, 6]. Moreover, the risk for developing psychopathology is high during adolescence and prodromal symptoms start even earlier and may overlap and are difficult to differentiate [5-8]. This has turned efforts towards identification and treatment of individuals at early stages of the illness, when first clinical manifestations emerge [8, 9].

Importantly, subthreshold symptoms of mania and depression along with unspecific behavioural, emotional, and cognitive manifestations are highly predictive of future manic and depressive episodes in BD as well as anxiety disorders, which is confirmed by the clinical staging perspective [10, 11]. Nevertheless, early recognition and intervention during the prodromal phase is still at an early stage in Sz [12] with limited research into valid prodromal criteria for BP [13]. Retrospective studies combining subjects with early-onset mania and early-onset first-episode psychosis have reported a similar pattern of neurodevelopmental and psychopathological features predating the appearance of more specific prodromal symptoms in both disorders [14, 15]. Therefore, the substantial overlap of symptoms in the initial phases suggests that early identification programmes should be aimed at detecting both the pre-psychotic and the pre-manic phases of SZ and BP [16]

ELIGIBILITY:
Inclusion Criteria:

- 6_18 years IQ > 70 parents of schizophrenia & mood disorders .

Exclusion Criteria:

* age <6 or >18 IQ < 70 .

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: families with one or two parents with psychiatric disorder.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-20 (Estimated); Primary Completion 2027-05-20 (Estimated); Study Completion 2027-08-20 (Estimated)

PRIMARY OUTCOMES:
Early recognition of psychiatric disorders among children and adolescents , So Early interventions to decrease the severity of the disorder can be done | 6 months
  Early recognition and intervention during the prodromal phase is still at an early stage in Sz [12] with limited research into valid prodromal criteria for BP [13]. Retrospective studies combining subjects with early-onset mania and early-onset first-episode psychosis have reported a similar pattern of neurodevelopmental and psychopathological features predating the appearance of more specific prodromal symptoms in both disorders [14, 15]. Therefore, the substantial overlap of symptoms in the initial phases suggests that early identification programmes should be aimed at detecting both the pre-psychotic and the pre-manic phases of SZ and BP [16].

SECONDARY OUTCOMES:
overlap of symptoms in the initial phases suggests that early identification | 6 months
  overlap of symptoms in the initial phases suggests that early identification programmes should be aimed at detecting both the pre-psychotic and the pre-manic phases of schizophrenia and bipolar disorders.

IPD SHARING:
Plan to Share IPD: No